CLINICAL TRIAL: NCT02611713
Title: DUOdopa/Duopa in Patients With Advanced Parkinson's Disease (PD) - a GLobal Observational Study Evaluating Long-Term Effectiveness (DUOGLOBE)
Brief Title: Observational Study Evaluating Long-Term Effectiveness of Duodopa/Duopa in Patients With Advanced Parkinson's Disease
Acronym: DUOGLOBE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-494
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Advanced Parkinson's Disease
Keywords: Advanced Parkinson's Disease; Duodopa/Duopa; carbidopa levodopa enteral suspension (CLES); levodopa-carbidopa intestinal gel (LCIG); OFF time; motor and non-motor symptoms; dyskinesia; tremor; Quality of Life; Observational; Long-term; Caregiver Burden; effectiveness; fluctuations
MeSH Terms: conditions — Dyskinesias; Tremor; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm A: Participants with Advanced Parkinson's Disease: Participants who along with their physicians have elected for treatment with Duodopa/Duopa and are prescribed according to the local product label and reimbursement guidelines for their participating countries.
- Arm B: Participants with Advanced Parkinson's Disease: Participants who along with their physicians have elected for treatment with Duodopa/Duopa and are prescribed according to the local product label and reimbursement guidelines for their participating countries. Participants will be evaluated with a wearable device

SUMMARY:
This study is a non-interventional post-marketing observational study (PMOS) of participants with advanced Parkinson's disease (PD) treated with Duodopa/Duopa in a routine clinical setting. Effectiveness of treatment will be collected with physician and participant/caregiver health outcomes beginning with PMOS enrollment (baseline visit), at the start of Duodopa/Duopa treatment via percutaneous endoscopic gastrostomy-with jejunal extension (PEG-J), at regularly scheduled visits closest to Months 3 and 6, and every 6 months thereafter up to 36 months. An additional cohort of participants will be enrolled who in addition will be evaluated with a wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for Duodopa/Duopa therapy in accordance with the approved local Duodopa/Duopa label in the participating country.
* Duodopa/Duopa naïve participants
* Decision to treat with Duodopa/Duopa made by the physician prior to any decision to approach the participant to participate in this study
* Prior to any study-related procedures being performed, the participant, or legal authorized representative (LAR) has voluntarily signed an Authorization for Use/Disclosure of Data (AUDD)/informed consent form (ICF) according to national regulations after the study has been explained and the subject has had the opportunity to have questions answered.
* For Arm B: Participant and caregiver must be motivated to use the PKG, understand the instructions and be able to handle the device.
* For Arm B: participant must demonstrate at least 75% concordance with the investigator's or qualified designee's assessment of symptoms on the Parkinson's disease diary following training at enrollment visit 1/V1 with concordance on at least 1 time interval of "Off", concordance on at least 1 time interval of "ON regardless of dyskinesia" and at least 1 time interval of "ON with dyskinesia" irrespective of whether the dyskinesia are troublesome or not troublesome.

Exclusion Criteria:

* Any condition included in the contraindications section of the approved local Duodopa/Duopa label in the participating country.
* Participants who have had previous surgery for PD including, but not limited to deep brain stimulation (DBS) or cell transplantation (this criterion removed for US sites for Arm A).
* Participants currently in treatment with continuous apomorphine infusion. In case of a previous treatment with continuous subcutaneous apomorphine infusion, there must be at least 4 weeks between discontinuation of this treatment and inclusion into this study.
* Mini-Mental State Examination (MMSE) score <24
* Participation in a concurrent interventional clinical trial.
* Lack of motivation or insufficient language skills to complete the study questionnaires

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Change in the number of hours spent in OFF time in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment on OFF time measured by the change (from baseline to 36 months) in the number of hours spent in OFF time as reported by the participant for the day prior to the clinical visit.
Change in Duration of OFF time (hours/day) in Arm B | Baseline visit (Enrollment) to month 6
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 6 months) in OFF time duration as measured by UPDRS Part IV (Motor Symptoms), item 39.
Change in Duration of OFF time (hours/day) in Arm B | Baseline visit (Enrollment) to month 6
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 6 months) in OFF time duration as reported by participant with PD Diary both per full 24 hours and for the time period of 09:00 - 18:00
Duration of bradykinesia score above target in Arm B | Baseline visit (Enrollment) to month 6
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 6 months) in duration of bradykinesia score above target between 09:00 - 18:00 and for the full 24 hours per day (measured by Parkinson's KinetiGraph ( PKG))
Average bradykinesia score in Arm B | Baseline visit (Enrollment) to month 6
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 6 months) in average bradykinesia score (measured by PKG)

SECONDARY OUTCOMES:
Change in Disease-Specific Caregiver Burden in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in disease-specific caregiver burden as measured by the Modified Caregiver Strain Index (MCSI) for PD with a total score range from 0 to 26.
Change in the Duration of Dyskinesia in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in duration of dyskinesia as reported by the patient for the day prior to the clinical visit
Change in Disease-Specific Sleep Quality in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in disease-specific sleep quality as measured by Parkinson's Disease Sleep Scale-2 (PDSS-2) with a total score range from 0 to 60.
Change in Tremor Severity in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in tremor severity as measured by UPDRS Part III, item 20 (Tremor at Rest) with a total score range of 0 to 20.
Change in Motor Function in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in motor function as measured by UPDRS, Part III (Motor Examination) with a total score range of 0 to 108.
Change in Generic Quality of Life in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in generic quality of life as measured by EuroQoL-5 Dimensions Quality of Life Questionnaire (EQ-5D). This assessment contains a health state descriptive part with five items scored from 1 to 3.
Change in Dyskinesia Severity in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in dyskinesia severity as measured by Unified Dyskinesia Rating Scale (UDysRS) with a total score range from 0 to 104.
Change in Overall Clinical Impression of Disease Severity in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in overall clinical impression of disease severity as measured by Clinical Impression of Severity Index for Parkinson's Disease (CISI-PD) obtained by adding four domain scores with a total score range from 0 to 24.
Change in Disease-Specific Quality of Life in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in disease-specific quality of life (QoL) as measured by Parkinson's Disease Questionnaire 8 (PDQ-8) summary index range from 0 to 100.
Change in OFF Time Duration in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in OFF time duration as measured by UPDRS Part IV (Motor Fluctuations), item 39, with a total score range of 0 to 4.
Change in Non-Motor Symptoms in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in non-motor symptoms as measured by Non-Motor Symptoms Scale (NMSS) with a total score range from 0 to 360.
Change in Healthcare Resource Utilization in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in healthcare resource utilization as measured by the Healthcare Resource Utilization Questionnaire (HCRU).
Change in Daytime Sleepiness in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in daytime sleepiness as measured by Epworth Sleepiness Scale (ESS) with a total score range from 0 to 24.
Change in Activities of Daily Living in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in Activities of Daily Living as measured by Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activity of Daily Living) with a total score range of 0 to 52.
Change in Complications of Therapy in Arm A | Baseline visit (Enrollment) to month 36
  Assess the effectiveness of Duodopa/Duopa treatment measured by the change (from baseline to 36 months) in Complications of Therapy (dyskinesia duration, disability, pain and early morning dystonia) as measured by UPDRS Part IV (Complications of Therapy), items 32 (individual score 0 to 4), 33 (individual score 0 to 4), 34 (individual score 0 to 4), 35 (individual score 0 to 1) and total score range of 0 to 13.
Correlation of non-motor and motor improvements with Quality of Life improvements in Arm A | Baseline visit (Enrollment) to month 36
  Assess the correlation of non-motor and motor improvements with the improvement in the Quality of Life (QOL).
Correlation between duration of OFF time measured by UPDRS IV and duration of bradykinesia score above target in Arm B | Baseline visit (Enrollment) to month 6
  Assess the correlation between duration of OFF time measured by UPDRS IV item 39 and duration of bradykinesia score above target between 09:00 - 18:00 and for the full 24 hours per day measured by PKG
Correlation between duration of OFF time measured by patient with PD Diary and average bradykinesia score in Arm B | Baseline visit (Enrollment) to month 6
  Assess the correlation between duration of OFF time measured by patient with PD Diary both per full 24 hours and for the time period of 09:00 - 18:00 and average bradykinesia score measured by PKG
Correlation between duration of bradykinesia score above target and average bradykinesia score in Arm B | Baseline visit (Enrollment) to month 6
  Assess the correlation between duration of bradykinesia score above target between 09:00 - 18:00 and for the full 24 hours per day measured by PKG and average bradykinesia score measured by PKG
Correlation between duration of OFF time measured by patient with PD Diary and duration of bradykinesia score above target in Arm B | Baseline visit (Enrollment) to month 6
  Assess the correlation between duration of OFF time measured by patient with PD Diary both per full 24 hours and for the time period of 09:00 - 18:00 and duration of bradykinesia score above target between 09:00 - 18:00 and for the full 24 hours per day measured by PKG
Correlation between duration of OFF time measured by UPDRS IV and average bradykinesia score in Arm B | Baseline visit (Enrollment) to month 6
  Assess the correlation between duration of OFF time measured by UPDRS IV item 39 and average bradykinesia score measured by PKG
Correlation between duration of dyskinesia and Unified Dyskinesia Rating Scale (UDysRS) in Arm B | Baseline visit (Enrollment) to month 6
  Pairwise correlation between duration of dyskinesia both per full 24 hours and 09:00 - 18:00 (based on UPDRS IV, PD diary and dyskinesia score measured by PKG) and UDysRS will be evaluated
Severity of dyskinesia in Arm B | Baseline visit (Enrollment) to month 6
  Severity of dyskinesia (item 33 score of UPDRS IV, UDysRS total score or the PKG-based dyskinesia score and the pairwise correlation between these will be evaluated
Motor symptoms in Arm B | Baseline visit (Enrollment) to month 6
  Motor symptoms measured by UPDRS III in ON state and correlation with PKG-based bradykinesia score will be evaluated
Severity of tremor in Arm B | Baseline visit (Enrollment) to month 6
  Severity of tremor measured by item 20 of UPDRS III in ON state and PKG-based tremor score and correlation between both will be evaluated
Activities of Daily Living (ADL) in Arm B | Baseline visit (Enrollment) to month 6
  ADL measured by UPDRS II in ON state and correlation with and PKG-based fluctuation/dyskinesia score and bradykinesia score will be evaluated
Sleep in Arm B | Baseline visit (Enrollment) to month 6
  Sleep as measured by PDSS-2, sleep/fatigue subdomain of NMSS, duration of sleep based on PD Diary or PKG-based night-time total sleep and pairwise correlation between these will be evaluated
Daytime sleepiness in Arm B | Baseline visit (Enrollment) to month 6
  Daytime sleepiness as measured by PKG-based percent of time asleep in the day time and the Epworth Sleepiness Scale and the correlation between these will be evaluated
Quality of Life (QoL) in Arm B | Baseline visit (Enrollment) to month 6
  QoL as measured by PDQ-8 and the correlation with PKG-based fluctuation/dyskinesia and bradykinesia scores will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (54):
- United States (19):
  - University of Alabama at Birmingham - Main /ID# 144422, Birmingham, Alabama
  - Parkinson's Disease and Moveme /ID# 144413, Boca Raton, Florida
  - University of Florida - Archer /ID# 144415, Gainesville, Florida
  - University of Miami /ID# 144420, Miami, Florida
  - Georgia Regents University /ID# 144417, Augusta, Georgia
  - University of Kansas Health Sy /ID# 154242, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center /ID# 144421, Lexington, Kentucky
  - Johns Hopkins University /ID# 144416, Baltimore, Maryland
  - Mercy St. Mary's Health Center /ID# 144418, Grand Rapids, Michigan
  - Jared Neuroscience Center /ID# 161629, Springfield, Missouri
  - Washington University-School of Medicine /ID# 147235, St Louis, Missouri
  - Univ Nebraska Med Ctr /ID# 147655, Omaha, Nebraska
  - Wake Forest Univ HS /ID# 144419, Winston-Salem, North Carolina
  - Penn State Child Hosp.Hersh,PA /ID# 160671, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 161135, Philadelphia, Pennsylvania
  - Vanderbilt Univ Med Ctr /ID# 150782, Nashville, Tennessee
  - University of Vermont Medical Center /ID# 144410, Burlington, Vermont
  - King County Public Hospital /ID# 144412, Kirkland, Washington
  - Northwest Neurological, PLLC /ID# 144409, Spokane, Washington
- Australia (4):
  - Concord Repatriation & Gen Hos /ID# 144373, Concord, New South Wales
  - St. Vincent's Hospital, Darlinghurst /ID# 144376, Darlinghurst, New South Wales
  - Kingston Centre /ID# 144374, Cheltenham, Victoria
  - Monash Medical Centre /ID# 144375, Clayton, Victoria
- Belgium (3):
  - UZ Antwerp /ID# 144378, Edegem
  - AZ Groeninge /ID# 144377, Kortrijk
  - CHU Tivoli /ID# 144379, La Louvière
- Hungary (2):
  - Semmelweis Egyetem /ID# 144381, Budapest
  - Pecsi Tudomanyegyetem Klinikai l.sz. Belgyogyaszati Klinika /ID# 144380, Pécs
- Israel (4):
  - Tel Aviv Sourasky Medical Center /ID# 153779, Tel Aviv, Tel Aviv
  - Assaf Harofeh Medical Center /ID# 144383, Be’er Ya‘aqov
  - The Edith Wolfson Medical Center /ID# 144382, Holon
  - Sheba Medical Center /ID# 147099, Ramat Gan
- Italy (3):
  - Ospedale Santo Stefano /ID# 144386, Prato
  - Azienda Ospedaliera Sant' Andrea /ID# 144385, Rome
  - A.O. Circolo e Fondazione Macc /ID# 144384, Varese
- Romania (7):
  - Institutul Clinic Fundeni /ID# 144448, Sector 2, București
  - Spitatlul Clinic Colentina /ID# 144447, Bucharest
  - Spital Universitar Bucuresti /ID# 144446, Bucharesti
  - Spitalul Clinic Judetean de Ur /ID# 144451, Oradea, Judet Bihor
  - Spitalul Clinic Judetean /ID# 144453, Târgu Mureş
  - Sp. Clinic de Judetean /ID# 144449, Timișoara
  - Sp. Clinic de Judetean /ID# 144452, Timișoara
- Univ Medical Ctr Ljubljana /ID# 144387, Ljubljana, Slovenia
- Spain (7):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 151782, Ferrol, A Coruna
  - Hospital Universitario Mutua Terrassa /ID# 144405, Terrassa, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 162277, Pamplona, Navarra, Comunidad
  - Hospital de Tortosa Verge de la Cinta /ID# 153502, Tortosa, Tarragona
  - OSI Ezkerraldea-Enkarterri-Cruces /ID# 151781, Barakaldo
  - Hospital Universitario Vall d'Hebron /ID# 151778, Barcelona
  - Hospital Universitario de Burgos /ID# 144406, Burgos
- United Kingdom (4):
  - King's College Hospital NHS /ID# 147130, London
  - St. George's Healthcare NHS /ID# 147131, London
  - Queens Hospital /ID# 147133, Romford
  - Salford Royal NHS Found Trust /ID# 151783, Salford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chaudhuri KR, Kovacs N, Pontieri FE, Aldred J, Bourgeois P, Davis TL, Cubo E, Anca-Herschkovitsch M, Iansek R, Siddiqui MS, Simu M, Bergmann L, Ballina M, Kukreja P, Ladhani O, Jia J, Standaert DG. Levodopa Carbidopa Intestinal Gel in Advanced Parkinson's Disease: DUOGLOBE Final 3-Year Results. J Parkinsons Dis. 2023;13(5):769-783. doi: 10.3233/JPD-225105. PMID 37302039
- [Derived] Aldred J, Anca-Herschkovitsch M, Antonini A, Bajenaru O, Bergmann L, Bourgeois P, Cubo E, Davis TL, Iansek R, Kovacs N, Kukreja P, Onuk K, Pontieri FE, Robieson W, Siddiqui MS, Simu M, Standaert DG, Chaudhuri KR. Application of the '5-2-1' screening criteria in advanced Parkinson's disease: interim analysis of DUOGLOBE. Neurodegener Dis Manag. 2020 Oct;10(5):309-323. doi: 10.2217/nmt-2020-0021. Epub 2020 Sep 2. PMID 32873195
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/search-results/?SearchTerm=NCT02611713&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&GenderDescriptions=&StudyTypes=STUDY_TYPE_OBSERVATIONAL&AttachmentTypes=&MileRadius=100&PageIndex=0&hasResults=&isHighValue=&SortField=&SortOrder=